CLINICAL TRIAL: NCT05616754
Title: Anhui Zhifei Longcom Biologic Pharmacy co. Ltd.
Brief Title: A Trial Evaluate the Immunogenicity and Safety of Recombinant COVID-19 Omicron-Delta Variant Vaccine (CHO Cell)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LKM-2022-NCV-GJ01
Record Dates: First submitted 2022-11-11; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: IgG; GMC
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group (Experimental): People more than 4 months after completing basic immunization with recombinant novel coronavirus protein vaccine (CHO cells)
  Interventions: Biological: Omicron-Delta Recombinant Novel Coronavirus Protein Vaccine (CHO cells)
- control group (Active Comparator): People more than 4 months after completing basic immunization with recombinant novel coronavirus protein vaccine (CHO cells)
  Interventions: Biological: Recombinant Novel Coronavirus Protein Vaccine (CHO cells)
- Observation group (Experimental): People over 4 months after completing basic immunization with COVID-19 mRNA vaccine
  Interventions: Biological: Omicron-Delta Recombinant Novel Coronavirus Protein Vaccine (CHO cells)

INTERVENTIONS:
Biological: Omicron-Delta Recombinant Novel Coronavirus Protein Vaccine (CHO cells) — The antigen protein of this product is designed to be expressed in tandem with Delta variant R319-N356 and Omicron variant R319-N356. The antigen is called DO-RBD for short.
  Arms: Observation group; Test group
Biological: Recombinant Novel Coronavirus Protein Vaccine (CHO cells) — This strain was made from the NCP-RBD receptor binding region of the spike glycoprotein of novel coronavirus expressed in recombinant CHO cells, which was purified and added with aluminum hydroxide adjuvant
  Arms: control group

SUMMARY:
The study was designed as a randomized, blind and controlled trial. A total of 300 patients aged 18 and above who were immunized with recombinant novel coronavirus protein vaccine (CHO cell) for more than 4 months (60 patients aged 60 and above) were randomly and blind divided into the experimental group and the control group, and received the experimental vaccine and the control vaccine, respectively.

In addition, 100 patients over 4 months after the completion of basic immunization with COVID-19 mRNA vaccine were selected as the open observation group, all of whom received 1 dose of experimental vaccine.

DETAILED DESCRIPTION:
The improved vaccine was developed against the Delta and Omicron COVID-19 variants. The overall design of this clinical trial was as follows: A total of 300 patients aged 18 and above who completed the basic immunization of recombinant novel coronavirus protein vaccine (CHO cell) for more than 4 months were randomly divided into the experimental group and the control group in a blind way, and were inoculated with the experimental vaccine and the control vaccine respectively. In addition, 100 patients over 4 months after the completion of basic immunization with COVID-19 mRNA vaccine were selected as the open observation group, all of whom received 1 dose of experimental vaccine. The main objective was to evaluate the immunogenicity and safety of Omicron-Delta recombinant novel coronavirus protein vaccine (CHO cells) against Omicron variants of novel coronavirus in people aged 18 years and above.

ELIGIBILITY:
Inclusion Criteria:

* Age eligible for observation in this clinical trial: adults aged 18 years and above
* Subjects voluntarily participate in this study, sign informed consent, provide legal identification, and understand and comply with the requirements of the test protocol
* More than 4 months after the completion of the whole course of recombinant novel coronavirus protein vaccine (CHO cell) basic immunization or more than 4 months after the completion of the novel coronavirus mRNA vaccine basic immunization
* Female and male participants of childbearing age took effective contraception during the study period

Exclusion Criteria:

* Prior history of severe allergy to any vaccine or to any component of the test vaccine, including aluminum preparation, such as anaphylactic shock, allergic laryngeal edema, purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), dyspnea, angineurotic edema, etc.;
* Suspected or confirmed fever (axillary temperature ≥37.3℃/ mouth temperature ≥37.5℃) within 72 hours before enrollment, or armpit temperature ≥37.3℃/ mouth temperature ≥37.5℃ on the day of enrollment;
* Confirmed cases of COVID-19 infection, asymptomatic infected persons or positive nucleic acid test history of COVID-19;
* Uncontrolled lymphoproliferative disease, unremission stage of aplastic anemia, active stage of primary immune thrombocytopenia (ITP), uncontrolled stage of coagulation disease, etc.
* a history of congenital or acquired immunodeficiency or autoimmune disease; Absence of spleen, or history of splenic surgery, trauma, or immunomodulator treatment within 6 months, such as immunosuppressive dose of glucocorticoids (dose reference: equivalent to prednisone 20mg/ day, over a week); Or monoclonal antibodies; Or thymosin; Or interferon; But topical use (such as ointments, eye drops, inhalants or nasal sprays) is permitted;
* Subunit vaccine and inactivated vaccine should be administered within 14 days before vaccination, and live attenuated vaccine should be administered within 30 days before vaccination;
* Patients with malignant tumors who are undergoing chemotherapy, radiotherapy or immunotherapy before and after surgery; Patients with organ transplant status;
* People with uncontrolled epilepsy and other progressive neurological diseases (e.g. Transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.);
* Patients with acute disease, or acute episodes of chronic disease, or uncontrolled severe chronic disease, such as medically uncontrolled hypertension (systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100mmHg);
* lactating or pregnant women;
* The investigator believes that the subject has any disease or condition that could put the subject at risk; The subject is unable to complete the trial as required by the protocol, and there are circumstances that interfere with the assessment of vaccine response.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Immunogenic end points | 6 months
  Geometric mean concentration (GMC) of RBD protein-binding Antibody (IgG) against Omicron variant of novel coronavirus at 14 days after vaccination in experimental group and control group.

SECONDARY OUTCOMES:
Immunogenic end points 2 | 6 months
  RBD protein-bound antibody (IgG) growth ratio (GMI) and positive turnover rate for Omicron variant of novel coronavirus at 14 days after vaccination in experimental group and control group;
Immunogenic end points 3 | 6 months
  RBD protein-binding antibody (IgG) GMC, GMI and positive turnover were detected against the primary COVID-19 strain and Delta variant 14 days after vaccination in experimental group.
Immunogenic end points 4 | 6 months
  RBD protein-binding antibody (IgG) GMC, GMI and positive turnover against the primary COVID-19 strain, Delta and Omicron variants 6 months after vaccination in the experimental group
Immunogenic end points 5 | 6 months
  RBD protein-binding antibody (IgG) GMC, GMI and positive turnover against the primary COVID-19 strain, Delta and Omicron variants were detected 14 days after vaccination in the observation group
Immunogenic end points 6 | 6 months
  RBD protein-binding antibody (IgG) GMC, GMI and positive turnover against the primary COVID-19 strain, Delta and Omicron variants in the observation group for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Erkin Musabaev, Dr., Principal Investigator — Research institute of virology
Locations (1):
- Uzbekistan, Tashkent city, Said baraka street 10, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li D, Duan M, Wang X, Gao P, Zhao X, Xu K, Gao GF. Neutralization of BQ.1, BQ.1.1, and XBB with RBD-Dimer Vaccines. N Engl J Med. 2023 Mar 23;388(12):1142-1145. doi: 10.1056/NEJMc2216233. Epub 2023 Mar 1. No abstract available. PMID 36856580